CLINICAL TRIAL: NCT02029716
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of RTA 408 Lotion in Healthy Volunteers
Brief Title: RTA 408 Lotion in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RTA 408-C-1305
Record Dates: First submitted 2013-12-30; First posted 2014-01-08 (Estimated); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: RTA 408; RTA 408 Lotion; Oxidative stress; Inflammation; Volunteers
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Part A (Placebo Comparator): RTA 408 lotion 0.5%, 1%, and 3% and lotion vehicle applied to skin twice daily for 14 days
  Interventions: Drug: RTA 408 Lotion 0.5%, 1%, 3%; Drug: Lotion vehicle/placebo
- Part B (Experimental): Up to 3% RTA 408 lotion applied to skin twice daily for 14 days (% concentration to be determined, based on results from Part A, ~100 cm2 surface area)
  Interventions: Drug: RTA 408 Lotion 0.5%, 1%, 3%
- Part C (Experimental): 3% RTA 408 lotion applied to skin twice daily for 28 days (~500 cm2 surface area)
  Interventions: Drug: RTA 408 Lotion 0.5%, 1%, 3%

INTERVENTIONS:
Drug: RTA 408 Lotion 0.5%, 1%, 3%
Drug: Lotion vehicle/placebo
  Arms: Part A

SUMMARY:
This study is a first-in-human study of a topical dermal lotion formulation of RTA 408, a novel small molecule which suppresses oxidative stress and inflammation. In this study, the safety, local pharmacodynamics (PD), and systemic pharmacokinetics (PK) of RTA 408 will be evaluated following topical application of RTA 408 Lotion to healthy volunteers. This study will be conducted in three parts. In Part A of the study, healthy volunteers will have RTA 408 Lotion Vehicle and RTA 408 Lotion (0.5%, 1%, and 3%) applied to a small skin surface area (four individual 4-cm2 sites; 16 cm2 total area) twice daily for 14 days to assess the local skin tolerability, local PD, and systemic PK of these treatments. Part B will be conducted after completion of Part A and will assess the safety, tolerability, local PD, and systemic PK of RTA 408 Lotion applied topically twice daily for 14 days to a larger skin surface area (~100 cm2). Part C will be conducted after completion of Part B and will assess the safety, tolerability, local PD, and systemic PK of RTA 408 Lotion applied topically twice daily for 28 days to a larger skin surface area (~500 cm2). The maximum tolerated drug concentration in Part A will be used in Part B and Part C.

Approximately 32 healthy adult volunteers will be enrolled in this study with 12 volunteers in Part A and 10 volunteers each, in Parts B and C.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must voluntarily give written informed consent and agree to comply with visit schedule including willingness to remain at the study site;
2. Subjects must be adults (male or female), ages 18 to 65, inclusive;
3. Subjects must have healthy skin on which reddening can easily be recognized (Fitzpatrick type I-IV skin);
4. The planned application site must have unbroken skin (ie, free from cuts, scratches, and abrasions), and be free of excessive hair, tattoos, or other abnormality that, in the Investigator's judgement, would interfere with the conduct of the study;
5. Subjects must have a body mass index (BMI) of ≥18 kg/m2 and ≤32 kg/m2;
6. Women must be of non-childbearing potential and may not be pregnant, lactating, or breast-feeding.
7. Male subjects must agree that they and any female partners will use 2 acceptable forms of contraception, 1 of which must be a condom, until 3 months after the last dose of study drug.

Exclusion Criteria:

1. Persons with Fitzpatrick skin types V or VI;
2. Presence of active inflammatory dermatoses (eg, atopic dermatitis, psoriasis), bacterial, viral, or fungal skin infections;
3. History of clinically significant drug allergies including allergies to any of the components of the investigational product and/or clinically significant food allergies as determined by the Investigator;
4. Use of any alcohol or methylxanthine-containing beverages or food (eg, coffee, tea, cola, chocolate, and "power drinks") from 72 hours prior to the first dose of study drug until after the last protocol specified blood sample;
5. Use of any tobacco products, nicotine-containing products, or pharmacologic smoking cessation therapy during the 3 months immediately prior to the first dose of study drug, and/or not willing or able to refrain from use of any of these products for the duration of the study until after the last protocol specified blood sample;
6. History of alcohol abuse within 2 years of the Screening Visit, in the judgment of the Investigator, or average weekly alcohol consumption of >14 alcoholic drinks. One drink is defined as 1 glass of beer (approximately 10 oz to 12 oz) or 1 can (12 oz) of beer, 1 glass of wine (approximately 4 oz to 5 oz), or 1 glass of distilled spirits (hard liquor) containing 1 oz of the liquor (1 oz of liquid is approximately 30 mL);
7. Positive breath test for alcohol at the Screening Visit or at Day -1;
8. History of drug abuse within 2 years of the Screening Visit, in the judgment of the Investigator;
9. Positive urine test for cotinine or drugs of abuse (ie, opiates, methadone, cocaine, amphetamines, cannabinoids, barbiturates, benzodiazepines) at the Screening Visit or at Day -1;
10. Not willing to abstain from strenuous exercise (eg, heavy lifting, weight training, calisthenics, aerobics) for at least 48 hours prior to admission to the investigational site until after the last protocol specified blood sample;
11. Use of substances known to be strong inhibitors or inducers of Cytochrome P450 (CYP450) enzymes (eg, ritonavir, ketoconazole, nefazodone, grapefruit juice) within 14 days prior to the first dose of study drug through the last study visit. Chronic exposure to enzyme inducers such as paint solvents or pesticides or other investigational drug use within 30 days prior to study drug administration;
12. Use of prescription drugs, dietary supplements, or herbal remedies (including products applied topically) within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study drug; use of non-prescription drugs or vitamins (including products applied topically) within 7 days prior to the first dose of study drug; or unwillingness to refrain from taking any such medication until after the last protocol specified blood sample;
13. Donation of whole blood >450 mL or blood products within 56 days prior to admission to the investigational site;
14. Use of any investigational drug within 30 days or 5 half-lives of the previous investigational drug prior to the first dose of study drug in this study, whichever is longer;
15. Positive screen for human immunodeficiency virus (HIV), hepatitis B, and/or hepatitis C at the Screening Visit;
16. Acute illness accompanied by temperature ≥101○F within 5 days prior to study drug administration;
17. Presence or history of cancer within 5 years prior to the Screening Visit (other than basal cell skin cancer in a location other than the back and without active lesions and adequately treated carcinoma in situ of cervix);
18. Presence or history of any significant cardiovascular, gastrointestinal, hepatic, renal, pulmonary, hematologic, endocrine, immunologic, dermatologic, neurologic disease
19. Presence of any other condition (including surgery) known to interfere with the absorption, distribution, metabolism, or excretion of medicines. History of appendectomy and cholecystectomy is permitted;
20. Any abnormal clinical laboratory value or abnormal electrocardiogram (ECG) finding at the Screening Visit or at Day -1 that is considered clinically significant by the Investigator;
21. International Normalized Ratio (INR) >1.5 at the Screening Visit;
22. Men whose female partner is pregnant or lactating, or who plans to become pregnant during the study or within 3 months after the end of the study;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2013-12-31 (Actual); Primary Completion 2014-04-01 (Actual); Study Completion 2014-04-01 (Actual)

PRIMARY OUTCOMES:
Skin changes or redness following topical application of RTA 408 lotion or lotion vehicle | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Medpace Clinical Pharmacology Unit, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Reisman SA, Goldsberry AR, Lee CY, O'Grady ML, Proksch JW, Ward KW, Meyer CJ. Topical application of RTA 408 lotion activates Nrf2 in human skin and is well-tolerated by healthy human volunteers. BMC Dermatol. 2015 Jul 14;15:10. doi: 10.1186/s12895-015-0029-7. PMID 26170027